CLINICAL TRIAL: NCT06981377
Title: Development of the PRIME Test for the Identification of Prostate Cancer Patients' Biomarkers Through Non-invasive Liquid Biopsies
Brief Title: PRostate Cancer Plasma Integrative Multi-modal Evaluation
Acronym: PRIME
Status: Recruiting | Type: Observational
Sponsor: Santa Chiara Hospital (Other)
Collaborators: Università degli Studi di Trento (Other)
Responsible Party: Principal Investigator, Orazio Caffo, Director, Medical Oncology Unit, Santa Chiara Hospital
Other Study IDs: PRIME - AA Trento
Record Dates: First submitted 2025-01-14; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Liquid biopsy; Cell free DNA (cfDNA); Extracellular Vesicles (EVs); Biomarkers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — DNA, B-Form

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat:
  * plasma is used for the isolation of cell free DNA (cfDNA) and extracellular Vesicles (EVs);
  * buffy coat is used for the extraction of genomic DNA (gDNA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metastatic Castration Resistant Prostate Cancer (mCRPC) patients: This group includes mCRPC patients treated with serial lines of treatment.
  For each line of treatment, blood samples are collected:
  1. Before starting the treatment;
  2. After 12 weeks;
  3. At the end of the treatment/progression.
  Interventions: Diagnostic Test: Analysis of cell free DNA, and extracellular vesicles (EVs) and EV-associated molecular components (including RNA, DNA, proteins)
- Metastatic Hormon Sensitive Prostate Cancer (mHSPC) patients: This group includes mHSPC patients treated with hormone therapy.
  In the hormone sensitive setting, blood samples are collected:
  1. Before starting the treatment;
  2. After 12 weeks;
  3. Every six months until progression to the castration resistant status.
  Interventions: Diagnostic Test: Analysis of cell free DNA, and extracellular vesicles (EVs) and EV-associated molecular components (including RNA, DNA, proteins)

INTERVENTIONS:
Diagnostic Test: Analysis of cell free DNA, and extracellular vesicles (EVs) and EV-associated molecular components (including RNA, DNA, proteins) — Plasma and buffy coat samples are shipped from the recruiting clinical sites to the lab of Professor Francesca Demichelis at the University of Trento (UniTN).
  At UniTN, samples are stored in dedicated freezers with restricted access and subsequently used as follows:
  * the plasma is used for the isolation of cell free DNA and extracellular vesicles (EVs);
  * the buffy coat is used for the extraction of genomic DNA.
  Nucleic acids sequencing library preparations and all downstream omics analyses are performed by Prof. Demichelis team.

SUMMARY:
The study aims to develop PRIME (PRostate cancer plasma Integrative Multi-modal Evaluation) liquid biopsy test and to implement its use to query prospectively collected samples in advanced prostate cancer (PCa) clinical trials and/or clinical settings. In order to maximise the utility of liquid biopsies for advanced PCa, PRIME is focused on the development of novel computational and sequencing approaches that integrate multiple information from plasma circulating elements: i) cell free DNA (cfDNA) gene mutation data with accurate quantitation of cfDNA structural genomic changes, ii) cfDNA genomic profiling with cfDNA methylation status, and iii) the information provided by extracellular vesicles (EVs) and EV-associated cargo (including DNA, RNA and proteins).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer
* Eligible for prostate cancer pharmacological treatment
* Given consent to study participation

Exclusion Criteria:

- Histological diagnosis other than prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected at oncology care clinics at participating clinical sites.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of circulating tumor DNA (ctDNA) in the plasma | From enrolment across different lines of treatment
  Number of circulating tumor DNA (ctDNA) in the plasma
Quantification of the fraction of cfDNA hypo/hypermethylation | From enrolment across different lines of treatment
  Rate of cfDNA hypo/hypermethylation
Presence of recurrent somatic aberrations in ctDNA (such as loss of RB1, TP53, BRCA1/2, or AR amplification). | From enrolment across different lines of treatment
  Assessment (yes/no) of recurrent somatic aberrations in ctDNA (such as loss of RB1, TP53,
Presence of Copy Number Variants (CNVs) in ctDNA | From enrolment across different lines of treatment
  Assessment (yes/no) of Copy Number Variants (CNVs) in ctDNA
Identification of EV-associated biomarkers | From enrolment across different lines of treatment
  Assessment (yes/no) of EV-associated biomarkers

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Istituto Romagnolo per lo Studio dei Tumori, Meldola, Forlì-Cesena
  - Azienda Ospedaliera San Luigi, Orbassano, Torino
  - Istituto Oncologico Veneto, Padua
  - Santa Chiara Hospital, Trento

REFERENCES:
- [Background] Mugoni V, Ciani Y, Quaini O, Tomasini S, Notarangelo M, Vannuccini F, Marinelli A, Leonardi E, Pontalti S, Martinelli A, Rossetto D, Pesce I, Mansy SS, Barbareschi M, Ferro A, Caffo O, Attard G, Di Vizio D, D'Agostino VG, Nardella C, Demichelis F. Integrating extracellular vesicle and circulating cell-free DNA analysis using a single plasma aliquot improves the detection of HER2 positivity in breast cancer patients. J Extracell Biol. 2023 Sep;2(9):e108. doi: 10.1002/jex2.108. Epub 2023 Sep 25. PMID 38046436
- [Background] Orlando F, Romanel A, Trujillo B, Sigouros M, Wetterskog D, Quaini O, Leone G, Xiang JZ, Wingate A, Tagawa S, Jayaram A, Linch M; PEACE Consortium; Jamal-Hanjani M, Swanton C, Rubin MA, Wyatt AW, Beltran H, Attard G, Demichelis F. Allele-informed copy number evaluation of plasma DNA samples from metastatic prostate cancer patients: the PCF_SELECT consortium assay. NAR Cancer. 2022 May 27;4(2):zcac016. doi: 10.1093/narcan/zcac016. eCollection 2022 Jun. PMID 35664542
- [Background] Conteduca V, Scarpi E, Wetterskog D, Brighi N, Ferroni F, Rossi A, Romanel A, Gurioli G, Bleve S, Gianni C, Schepisi G, Lolli C, Cortesi P, Matteucci F, Barone D, Paganelli G, Demichelis F, Beltran H, Attard G, De Giorgi U. Plasma tumor DNA is associated with increased risk of venous thromboembolism in metastatic castration-resistant cancer patients. Int J Cancer. 2022 Apr 1;150(7):1166-1173. doi: 10.1002/ijc.33834. Epub 2021 Oct 13. PMID 34605002
- [Background] Conteduca V, Wetterskog D, Scarpi E, Romanel A, Gurioli G, Jayaram A, Lolli C, Tandefelt DG, Schepisi G, Casadei C, Wingate A, Matteucci F, Paganelli G, Gonzalez-Billalabeitia E, Demichelis F, De Giorgi U, Attard G. Plasma tumour DNA as an early indicator of treatment response in metastatic castration-resistant prostate cancer. Br J Cancer. 2020 Sep;123(6):982-987. doi: 10.1038/s41416-020-0969-5. Epub 2020 Jul 16. PMID 32669676
- [Background] Wu A, Cremaschi P, Wetterskog D, Conteduca V, Franceschini GM, Kleftogiannis D, Jayaram A, Sandhu S, Wong SQ, Benelli M, Salvi S, Gurioli G, Feber A, Pereira MB, Wingate AM, Gonzalez-Billalebeitia E, De Giorgi U, Demichelis F, Lise S, Attard G. Genome-wide plasma DNA methylation features of metastatic prostate cancer. J Clin Invest. 2020 Apr 1;130(4):1991-2000. doi: 10.1172/JCI130887. PMID 32149736
- [Background] Beltran H, Romanel A, Conteduca V, Casiraghi N, Sigouros M, Franceschini GM, Orlando F, Fedrizzi T, Ku SY, Dann E, Alonso A, Mosquera JM, Sboner A, Xiang J, Elemento O, Nanus DM, Tagawa ST, Benelli M, Demichelis F. Circulating tumor DNA profile recognizes transformation to castration-resistant neuroendocrine prostate cancer. J Clin Invest. 2020 Apr 1;130(4):1653-1668. doi: 10.1172/JCI131041. PMID 32091413
- [Background] Prandi D, Demichelis F. Ploidy- and Purity-Adjusted Allele-Specific DNA Analysis Using CLONETv2. Curr Protoc Bioinformatics. 2019 Sep;67(1):e81. doi: 10.1002/cpbi.81. PMID 31524989
- [Background] Vagner T, Spinelli C, Minciacchi VR, Balaj L, Zandian M, Conley A, Zijlstra A, Freeman MR, Demichelis F, De S, Posadas EM, Tanaka H, Di Vizio D. Large extracellular vesicles carry most of the tumour DNA circulating in prostate cancer patient plasma. J Extracell Vesicles. 2018 Aug 7;7(1):1505403. doi: 10.1080/20013078.2018.1505403. eCollection 2018. PMID 30108686
- [Background] Romanel A, Gasi Tandefelt D, Conteduca V, Jayaram A, Casiraghi N, Wetterskog D, Salvi S, Amadori D, Zafeiriou Z, Rescigno P, Bianchini D, Gurioli G, Casadio V, Carreira S, Goodall J, Wingate A, Ferraldeschi R, Tunariu N, Flohr P, De Giorgi U, de Bono JS, Demichelis F, Attard G. Plasma AR and abiraterone-resistant prostate cancer. Sci Transl Med. 2015 Nov 4;7(312):312re10. doi: 10.1126/scitranslmed.aac9511. PMID 26537258
- [Background] Carreira S, Romanel A, Goodall J, Grist E, Ferraldeschi R, Miranda S, Prandi D, Lorente D, Frenel JS, Pezaro C, Omlin A, Rodrigues DN, Flohr P, Tunariu N, S de Bono J, Demichelis F, Attard G. Tumor clone dynamics in lethal prostate cancer. Sci Transl Med. 2014 Sep 17;6(254):254ra125. doi: 10.1126/scitranslmed.3009448. PMID 25232177
- [Background] Prandi D, Baca SC, Romanel A, Barbieri CE, Mosquera JM, Fontugne J, Beltran H, Sboner A, Garraway LA, Rubin MA, Demichelis F. Unraveling the clonal hierarchy of somatic genomic aberrations. Genome Biol. 2014 Aug 26;15(8):439. doi: 10.1186/s13059-014-0439-6. PMID 25160065
- [Result] Franceschini GM, Quaini O, Mizuno K, Orlando F, Ciani Y, Ku SY, Sigouros M, Rothmann E, Alonso A, Benelli M, Nardella C, Auh J, Freeman D, Hanratty B, Adil M, Elemento O, Tagawa ST, Feng FY, Caffo O, Buttigliero C, Basso U, Nelson PS, Corey E, Haffner MC, Attard G, Aparicio A, Demichelis F, Beltran H. Noninvasive Detection of Neuroendocrine Prostate Cancer through Targeted Cell-free DNA Methylation. Cancer Discov. 2024 Mar 1;14(3):424-445. doi: 10.1158/2159-8290.CD-23-0754. PMID 38197680